CLINICAL TRIAL: NCT02771379
Title: A Non-interventional Study of Clinical Experience in Patients Prescribed Raxone® for the Treatment of Leber's Hereditary Optic Neuropathy (LHON)
Brief Title: Post Authorisation Safety Study With Raxone in LHON Patients
Acronym: PAROS
Status: Completed | Type: Observational
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNT-IV-003
Record Dates: First submitted 2016-04-25; First posted 2016-05-13 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Leber's Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — idebenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients who are treated with Raxone®
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Idebenone — Raxone 900mg/day as per Raxone SmPC and medical judgement of treating physician.
  Other Names: Raxone®

SUMMARY:
This study is a multicentre, prospective, non-interventional post-authorisation safety study (PASS) of the clinical outcomes for patients with LHON treated with Raxone®.

No medication will be provided as part of this study. Raxone® will be obtained through commercial channels.

ELIGIBILITY:
Inclusion Criteria:

* Patient prescribed Raxone® for the treatment of LHON;
* Patient has completed an Informed Consent Form (ICF) indicating that he/she (or a legally acceptable representative) has been informed of all pertinent aspects of the study and has agreed to participate in the study;
* Patient is not participating in any interventional study.

Exclusion Criteria:

* No explicit exclusion criteria exist to avoid selection bias and to allow for documentation of routine clinical practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient prescribed Raxone® for the treatment of LHON who have completed the informed consent. This study will be conducted in EU in approximately 45 highly specialized centres in ophthalmology and neuroophthalmology.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2016-09; Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Long-term safety profile of Raxone® in the treatment of patients with LHON when used under conditions of routine clinical care. | up to 5 years
  Safety will be assessed by the collection and analysis of adverse events of special interest (AESIs), frequency and nature of AEs and serious adverse events (SAEs), adverse drug reactions (ADRs) and serious adverse drug reactions (SADRs)

SECONDARY OUTCOMES:
Long-term effectiveness of Raxone® in the treatment of patients with LHON when used under conditions of routine clinical care | up to 5 years
  According to the Summary of Product Characteristics (SmPC) a patient's vision should be continually monitored therefore effectiveness will be assessed by measuring on-therapy changes in patients' visual acuity (VA), visual fields (VF), colour contrast sensitivity and Retinal Nerve Fibre Layer thickness (RNFL) where available.

CONTACTS AND LOCATIONS:
Locations (26):
- Austria (2):
  - Universitaetsklinikum Graz, Graz
  - Medical University of Vienna, Vienna
- France (9):
  - CHU de Nîmes - Hôpital Carémeau, Nîmes, Gard
  - CHU Angers - Hôpital Hôtel Dieu, Angers, Maine Et Loire
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital Européen Georges Pompidou, Paris, Paris Cedex 15
  - CHU Amiens - Centre Saint Victor, Amiens, Somme
  - Hospices Civils de Lyon, Lyon
  - Hopital Neurologique Pierre Wertheimer, Lyon
  - Centre Hospitalier National d'Ophtalmologie (CHNO) des Quinze-Vingts, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
- Germany (9):
  - Julius Maximilians University, Würzburg, Bavaria
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Friedrich-Baur-Institut, Munich
  - Universitaetsklinikum Muenster, Münster
  - Dietrich-Bonhoeffer-Klinikum Neubrandenburg, Neubrandenburg
  - Universitaetsklinikum Regensburg, Regensburg
- Athens Ophthalmological Center, Athens, Greece
- Italy (3):
  - Università di Bologna-Clinica Neurologica-Dipartimento di Scienze Neurologiche, Bologna
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera S. Camillo Forlanini, Rome
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht University Medical Center, Maastricht